CLINICAL TRIAL: NCT01345526
Title: A Double Blind Placebo Controlled Randomized Phase II Study Evaluating the Efficacy and Safety of the Prophylactic Use of Doxycycline +/- Vitamin K Cream in First Line mCRC Patients Treated With Erbitux and FOLFIRI.
Brief Title: Efficacy and Safety of the Prophylactic Use of Doxycycline +/- Vitamin K Cream
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Universitätsmedizin Mannheim (Other)
Responsible Party: Principal Investigator, Ralf Hofheinz, Head TTZ University Hospital Mannheim, Universitätsmedizin Mannheim
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Supportive Care
Other Study IDs: E-VITA
Record Dates: First submitted 2011-04-21; First posted 2011-05-02 (Estimated); Last update posted 2021-04-30 (Actual); Status verified 2011-04

CONDITIONS: Metastatic Colorectal Cancer
MeSH Terms: conditions — Colorectal Neoplasms

STUDY DESIGN:
Intervention Model Description: Randomized Phase II trial
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Randomized Phase II Trial assessing the prevention of acne like Skin rash
Oversight: Data Monitoring Committee: No

ARMS (2):
- Metastatic colorectal cancer, Doxycycline, Vitamin K1 Cream (Experimental)
  Interventions: Device: Reconval K1 Cream
- Metastatic colorectal cancer, Doxycycline, Cream (Placebo Comparator)
  Interventions: Device: Reconval Cream

INTERVENTIONS:
Device: Reconval K1 Cream
  Arms: Metastatic colorectal cancer, Doxycycline, Vitamin K1 Cream
Device: Reconval Cream
  Arms: Metastatic colorectal cancer, Doxycycline, Cream

SUMMARY:
The aim of this Phase 2, two-arm, randomized, double blind placebo controlled study is to evaluate the efficacy of combination therapy of doxycycline and Vitamin K1 compared to doxycycline plus placebo for the prevention of acne-like skin rash in mCRC patients receiving first line cetuximab treatment.

DETAILED DESCRIPTION:
The aim of this Phase 2, two-arm, randomized, double blind placebo controlled study is to evaluate the efficacy of combination therapy of doxycycline and Vitamin K1 compared to doxycycline plus placebo for the prevention of acne-like skin rash in mCRC patients receiving first line cetuximab treatment.

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent must be given
* Patient ≥ 18 years
* Histologically proven and measurable metastatic adenocarcinoma of the colon or rectum (according to modified RECIST criteria v.1.1)
* Patients eligible for Erbitux and FOLFIRI treatment K-Ras wild type tumour
* Metastatic disease
* Life expectancy of at least 12 weeks
* WHO performance status of 0 or 1
* Effective contraception for both male and female patients if the risk of conception exists
* Adequate organ function
* Adequate bone marrow, hepatic and renal function (Hemoglobin > 10.0 g/dL, platelet count > 100 x 109/L, absolute neutrophil count > 1.5 x 109/L; ALAT, ASAT < 2.5 x ULN (upper limit of normal range) or < 5x ULN in case of liver metastasis; Alkaline phosphatase < 2.5 x ULN; Total bilirubin < 1.5 x ULN; Creatinine clearance > 50 mL/min (calculated according to Cockcroft and Gault formula)).

Exclusion Criteria:

* Prior treatment for metastatic disease (adjuvant therapy with 5-FU/oxaliplatin based regimens) allowed if stopped 6 months prior to registration on study
* Prior treatment with EGFR inhibitor
* Surgery (excluding diagnostic biopsy) or irradiation within 4 weeks prior to study entry
* Administration of any investigational drug or agent/procedure, i.e. participation in another trial within 4 weeks before beginning treatment with study drugs
* Concurrent chronic systemic immune therapy, chemotherapy, radiation therapy or hormone therapy not indicated in the study protocol
* Any active dermatological condition > grade 1 at baseline possibly interfering with or influencing the results or conduct of the present study
* Brain metastasis (known or suspected)
* Significant impairment of intestinal resorption (e.g. chronic diarrhea, inflammatory bowel disease)
* Any other uncontrolled concomitant illness, including serious uncontrolled intercurrent infection
* Severe or uncontrolled cardiovascular disease (congestive heart failure NYHA III or IV, unstable angina pectoris, history of myocardial infarction within the last twelve months, significant arrhythmias)
* Known allergy or any other adverse reaction to any of the study drugs or to any related compound.
* Any organ allograft requiring immunosuppressive therapy.
* Pregnancy (absence to be confirmed by serum/urine beta human chorion gonadotrophin (HCG)) or breast-feeding.
* Other previous malignancy within 5 years, with exception of a history of a previous basal cell carcinoma of the skin or pre-invasive carcinoma of the cervix surgically cured or adequately treated.
* Known drug abuse / alcohol abuse
* Legal incapacity or limited legal capacity
* Any psychological, familial, sociological or geographical condition potentially hampering compliance with the study protocol and followup schedule; those conditions should be discussed with the patient before registration in the trial.
* Medical or psychological condition which, in the opinion of the investigator, would not permit the patient to complete the study or meaningfully sign informed consent.
* Known M. Meulengracht (Gilbert´s disease) or DPD-insufficiency
* Known coagulation disorders
* Ongoing or planned treatment with coumarin derivates

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 124 (Actual)
Dates: Start 2011-04; Primary Completion 2016-12 (Actual); Study Completion 2016-12 (Actual)

PRIMARY OUTCOMES:
Occurrence of acne-like skin rash grade ≥ 2 (according to the CTCAE) version 4.02) during the 8 weeks of skin treatment. | Week 8
PFS rate, toxicity, compliance | Week 8

CONTACTS AND LOCATIONS:
Overall Officials: Ralf Hofheinz, Prof., Study Chair — Universitätsmedizin Mannheim
Locations (2):
- Unversity Hospital Mannheim, Mannheim, Germany
- Institute of Oncology Ljubljana, Ljubljana, Slovenia